CLINICAL TRIAL: NCT04087642
Title: CREDE Study: Intraoperative Crede Manoeuver Compared to Preoperative Prolapse Reduction Stress Test to Predict Postoperative de Novo Stress Urinary Incontinence (PONSUI) at the Time of Pelvic Organ Prolapse (POP) Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: St. Mary's Research Centre, Montreal (Unknown)
Responsible Party: Principal Investigator, Maryse Larouche, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MP-37-2019-4845
Record Dates: First submitted 2019-09-04; First posted 2019-09-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Pelvic Organ Prolapse; de Novo Stress Urinary Incontinence; Stress Urinary Incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoperative Crede manoeuver (Experimental): Method 1 (M1) consists in intraoperative Crede maneuver: After POP surgical reduction, the bladder will be retrograde filled with 300 ml of sterile water through a catheter that will then be removed. Brief and forceful suprapubic pressure will be applied. The test is positive if the surgeon visualizes a urinary leak.
  In this group, the intraoperative Crede manoeuver will determine if an anti-incontinence procedure should be performed concomitantly.
  Interventions: Diagnostic Test: Intraoperative Crede manoeuver
- Preoperative prolapse reduction cough stress test (Active Comparator): An examiner will perform the test preoperatively in the office, at the same visit as the recruitment. With a volume of 250-350 mL of urine in the bladder (confirmed by bladder scanner), a prolapse reduction cough stress test will be performed (posterior speculum blade for reduction). The test is positive if the examiner visualizes a urinary leak.
  In this group, the preoperative prolapse reduction cough stress test will determine if an anti-incontinence procedure should be performed concomitantly.
  Interventions: Diagnostic Test: Preoperative prolapse reduction cough stress test

INTERVENTIONS:
Diagnostic Test: Intraoperative Crede manoeuver — In this group, both tests will be performed but the intraoperative Crede manoeuver will determine if an anti-incontinence procedure should be performed concomitantly. If the test is positive, it will be performed. If the test is negative, it will not be performed.
  Arms: Intraoperative Crede manoeuver
Diagnostic Test: Preoperative prolapse reduction cough stress test — In this group, both tests will be performed but the preoperative prolapse reduction cough stress test will determine if an anti-incontinence procedure should be performed concomitantly. If the test is positive, it will be performed. If the test is negative, it will not be performed.
  Arms: Preoperative prolapse reduction cough stress test

SUMMARY:
The CREDE pilot randomized study will compare the intraoperative Crede manoeuver (M1) to preoperative prolapse (POP) reduction cough stress test (M2) for the prediction and prevention of PONSUI. The rates of PONSUI and its effect on patient reported outcomes and quality of life will be determined among women with positive or negative tests, and those with and without concomitant anti-incontinence procedure performed. This information will help inform larger studies on the topic.

DETAILED DESCRIPTION:
Primary objective

* To assess feasibility of a pilot study to test this hypothesis with the goal to conduct a full trial (sample size calculation, validation of instruments used, randomization processes)
* To estimate the rate of subjective PONSUI at 6 weeks and at 6 months in continent women undergoing POP surgical repair where a positive intraoperative Crede maneuver (M1) vs. a positive preoperative prolapse reduction stress test (M2) are used to select candidates for concomitant anti-incontinence procedure (either 1. retropubic midurethral sling (MUS) or 2. periurethral bulking injections)

Secondary objectives

I. To compare the estimated rate of objective PONSUI at 6 weeks and at 6 months (as determined by cough stress test) in continent women undergoing POP surgical repair where a positive intraoperative Crede maneuver (M1) vs. a positive preoperative prolapse reduction stress test (M2) are used to select candidates for concomitant anti-incontinence procedure II. To compare the rate of urinary symptoms and the effect on quality of life at 6 weeks and 6 months between M1 and M2, by Urinary Distress Inventory (UDI-6) and Urinary Impact Questionnaire (UIQ-7) III. To describe the risk of complications in patients having either maneuvers (M1, M2), including bladder perforation, voiding dysfunction, urinary tract infection and mesh exposure IV. To assess the concordance/discordance rate of M1 and M2 to compare the predictive subjective and objective PONSUI values of both maneuvers by test results and by anti-incontinence procedure

Methodology

This is a pilot randomized controlled study of two parallel groups, in a sample of 110 continent women undergoing surgical correction of symptomatic pelvic organ prolapse (POP). The sample will be drawn from women presenting to three urogynecologists at St-Mary's hospital and McGill University Health Center (MUHC).

Intervention:

The patients will be randomized in two groups, allocated in a 1:1 ratio. All participants will undergo both methods to evaluate their risk of PONSUI. Method 1 (M1) consists in intraoperative Crede maneuver. Method 2 (M2) consists in a preoperative prolapse reduction stress test. In group A: A positive M1 will determine performance of anti-incontinence procedure. In group B: A positive M2 will determine performance of anti-incontinence procedure.

Surgical Procedure In both groups, women will have their planned surgery for POP correction under spinal (regional) or general anesthesia. The POP repair followed by the M1 will be performed for all women. The result of preoperative M2 won't be available to surgeon at the moment of performing M1. If the PONSUI prediction test for which the patient had been randomized to is positive, we will perform the anti-incontinence procedure selected by the patient (1. retropubic midurethral sling (MUS), or 2. periurethral bulking injections) after the POP repair. Placement of MUS and periurethral bulking injections will follow standardized reported technique. After the surgical procedure, a Foley catheter or suprapubic catheter will be inserted, and removed on postoperative day one. After catheter removal, a trial of void protocol is in place at our institutions. If post void residual volume by bladder scanner is over 250 mL, the Foley catheter will be reinserted and left in place for one week (or the suprapubic catheter will be kept for one week), while prophylactic antibiotics are given.

Randomization:

To address potential imbalances across study groups a computer-generated (SAS version 9.4) randomization schedule will be stratified by surgeon (3-5 different surgeons) and type of incontinence procedure chose (1. MUS, 2. Bulking), using random block sizes of 2 or 4, with an allocation ratio of 1:1. In order to ensure allocation concealment, the research assistant will first verify eligibility and informed consent, and then assign a study ID to each participant. Prior to the surgical procedure, the research assistant will enter this information plus the surgeon and incontinence procedure type into an automated interface prepared by the statistician. The result of randomization will be available to the surgeon only in the operating room (OR), after both the preoperative M2 and the intraoperative M1 have been performed. Specifically, the primary surgeon will be blinded until immediately after the M1 is performed and the result is recorded. The research assistant will have left an envelope with the randomization group in the OR prior to the beginning of the procedure. This envelope will be opened after the M1 is performed. The result of M2 will also be available if the woman is randomized to group B.

Sample size consideration:

Approximately 200 patients undergo POP surgical repair surgery per year in the two centers where the study will be conducted. For the pilot study, we are planning to recruit 100 eligible patients (50 per group) into the study with an added 10% estimated dropout rate for an overall total of 110 patients (55 per group). To the best of our knowledge, no previous study exists which would allow us to perform the appropriate sample size calculations. To do so, we would need some estimate of the rate of subjective PONSUI after intraoperative Crede maneuver (M1) at 6 weeks and 6 months. It is one of the purposes of this pilot project to determine such a parameter for planning a future randomized controlled trial. The rate of subjective PONSUI after preoperative prolapse reduction stress test (M2) varies around 14%, 54%, 17%, 26% for positive tests with and without anti-incontinence surgery and for negative tests with and without anti-incontinence surgery respectively. We thus estimate an overall rate of 30% PONSUI with the use of the preoperative prolapse reduction stress test. In the absence of an educated guess, we have verified that with our sample size (50 in each group) the minimal significant difference of 22% (30% vs 8%) between two groups PONSUI rates could be detected with a power of at least 80% using Pearson chi-squared and a confidence level of α = 0.05. Also, a set of relevant baseline imbalances will be pre-specified (recruitment site and prolapse stage "II vs III-IV") and a stratified randomization will be performed.

Data gathering Variables collected will include age, medication (including hormonal therapy), smoking status, diabetes, past obstetrical history (including parity, vaginal deliveries and cesarean sections), previous surgery for POP (type), previous hysterectomy, menopausal status, daytime frequency and nocturia. Patient will also answer validated questionnaires on urinary symptoms and impact on quality of life including: 1. Urinary Distress Inventory (UDI-6), and 2. Urinary Impact Questionnaire (UIQ-7).

At baseline, physical examination will be performed by one of the three participating urogynecologists or one of the urogynecology fellows. It will include POP-Q evaluation, genitourinary atrophy assessment, myofascial pain (pain at palpation of the vaginal muscles), and the preoperative prolapse reduction stress test (M2) for all women (positive/negative). After the exam, women will be asked to urinate and we will estimate the post void residual volume (urine left into the bladder after a micturition) with a bladder scanner.

At the moment of the surgery to correct the POP, all of the women will have a Crede maneuver assessment (M1). The result of the test will be noted (positive/negative). Information collected at the time of the surgery will include date, type of surgery, type of anesthesia (general or regional), estimated blood loss, perioperative complications (as bladder and urethral perforation or hemorrhage). Postoperative complications such as postoperative urinary retention (use of Foley/suprapubic catheter for seven days or more), and urinary tract infection will also be recorded.

Women will follow the usual postoperative visit calendar used in our institutions (visit 6 weeks and 6 months after the surgery). They will fill the same two questionnaires (UDI-6 and UIQ-7) that they answered at the beginning of the study. A blinded urogynecologist or a fellow in urogynecology will perform an examination. The amount of urine into the bladder will be estimated with a bladder scanner. A cough stress test will be done with an amount estimated between 250-350 mL of urine. The patient will be asked to drink water if the bladder is not full enough. The women have to cough strongly while in supine position. The examiner will note if he sees urine leakage (positive test) or not (negative test). He/she will also do a vaginal examination to note prolapse stage (POP-Q), and if there are any complication including mesh erosion or extrusion and important pain.

The research assistant will be involved at the time of women's recruitment, to ensure patient randomization, to coordinate postoperative examinations by a blinded examiner, and for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Anterior, uterine or apical prolapse with a POP-Q stage II or more requiring surgical correction

Exclusion Criteria:

* Stress urinary incontinence (SUI) on history
* Previous anti-incontinence surgery
* Pregnancy
* Prior urethral repair surgery (diverticulum, fistula)
* Women who do not speak or read English or French
* Isolated posterior compartment prolapse
* Geographic location preventing women to come to 6 week and 6 month appointments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Subjective postoperative de novo stress urinary incontinence (PONSUI) | 6 months
  SUI occurring after a surgery (usually a prolapse correction) in a patient who did not have SUI before the surgery. In this study, PONSUI is defined as answering "yes" to question #3 in the UDI-6 questionnaire: "Do you experience urine leakage related to activity, coughing or sneezing?" after the surgery, in previously continent women.

SECONDARY OUTCOMES:
Objective PONSUI | 6 months
  Positive cough stress test
Urinary symptoms | 6 months
  Scores on Urinary Distress Inventory (UDI-6)
Complications | 6 months
  Perioperative and postoperative complications including: bladder perforation, voiding dysfunction, urinary tract infection and mesh exposure
Prevalence and correlation of each test result | At baseline
  Percentage of positive tests and correlation between both tests
Impact on quality of life | 6 months
  Urinary Impact Questionnaire (UIQ-7)

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Larouche, MD, MPH, Principal Investigator — St. Mary's Research Centre and RI-MUHC
Locations (2):
- Canada (2):
  - St. Mary's Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No